CLINICAL TRIAL: NCT01488032
Title: Differences in Nerve Fiber Layer Between Patients With Normal- and High-Pressure-Glaucoma With Similar Structural Optic Nerve Damage
Brief Title: Differences in Nerve Fiber Layer Between Patients With Normal- and High-Pressure-Glaucoma
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Other Study IDs: EK 322102010
Record Dates: First submitted 2011-12-01; First posted 2011-12-08 (Estimated); Last update posted 2011-12-09 (Estimated); Status verified 2011-12

CONDITIONS: Normal Tension Glaucoma; High Tension Glaucoma
MeSH Terms: conditions — Low Tension Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- high-tension glaucoma: subjects with IOP>22 mmHg without eyedrops and signs of glaucomatous optic nerve damage
- low-tension glaucoma: subjects with IOP<22 mmHg without eyedrops and signs of glaucomatous optic nerve damage

SUMMARY:
The purpose of the study is to prove if there is any difference in the nerve fiber layer between patients with normal- and high-tension-glaucoma with similar structural optic nerve head parameters.

DETAILED DESCRIPTION:
It is till now not definitely clear whether normal- and high-tension glaucoma are different forms of the same disease and whether they have similar pathogenetic mechanisms. Spectral domain optical coherence tomography (SD-OCT) is supposed to objectively evaluate retinal nerve fiber layer (RNFL) thickness. The investigators propose a study to compare the RNFL in patients with normal- and high-tension-glaucoma. In order to exclude other possible differences,which could influence the results, only patients with similar structural optic nerve head damage in both groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* persons over 18 years
* men or women
* with normal- and high-tension glaucoma

Exclusion Criteria:

* cataract
* cloudy cornea and other conditions with bad visualisation quality of optic nerve head
* optic nerve atrophy except glaucomatous

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: primary care clinic University hospital of Dresden
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2011-03; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
RNFL in different segments | up to 9 Months
  RNFL in upper, lower, temporal and nasal segments